CLINICAL TRIAL: NCT03467828
Title: Investigation of Polymorphisms Defined in Specific Genes Which Are Associated With Bronchopulmonary Dysplasia In Turkish Population
Brief Title: Investigation of Polymorphisms in Bronchopulmonary Dysplasia In Turkish Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seda Yilmaz Semerci (Other)
Responsible Party: Sponsor-Investigator, Seda Yilmaz Semerci, Neonatologist, MD, Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 18
Record Dates: First submitted 2018-03-05; First posted 2018-03-16 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Bronchopulmonary Displasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Infants diagnosed with BPD.
  Interventions: Genetic: polymorphism analyzing
- Control Group (No Intervention): Infants born in similar gestational week and birth weight but not diagnosed with BPD.

INTERVENTIONS:
Genetic: polymorphism analyzing — Blood samples will be taken to EDTA containing tubes and then will be analyzed for genetic polymorphisms.
  Arms: Study Group

SUMMARY:
Bronchopulmonary dysplasia (BPD) is a chronic lung disease that affects a ratio of up to 20-30% of infants prematurely born before 30rd week. Delay of starting to speak, cerebral palsy and cognitive disorders may be seen in infants suffering from this disease. Although all the evidence found on the specific mediators and pathways that regulate the mechanism by studies made to understand the pathophysiologic mechanism, there hasn't been any remarkable progress on preventing the development of BPD in new-born infants born below 1500gr body weight. BPD is still one of the most important morbidity and mortality reasons in premature infants. There is a need of further studies to understand the genetic background of BPD specific to different populations, to identify polymorphisms related with the disease and for developing genetic methods for early the diagnose of the disease.

With this purpose, first of all polymorphisms related with BPD and those which are related with similar other lung diseases will be investigated. DNA samples derived from blood samples of 200 patients (100 BPD infant and 100 control) will be examined for polymorphisms in specific genes that are chosen in the light of the prior literature scanning. To the investigators' knowledge, this will be the first study of a broad scanning of polymorphisms related with BPD in Turkish population.

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia is a chronic lung disease that affects a ratio of up to 20-30% of infants prematurely born before 30rd week. Delay of starting to speak, cerebral palsy and cognitive disorders may be seen in infants suffering from this disease. Although all the evidence found on the specific mediators and pathways that regulate the mechanism by studies made to understand the pathophysiologic mechanism, there hasn't been any remarkable progress on preventing the development of BPD in new-born infants born below 1500gr body weight. BPD is still one of the most important morbidity and mortality reasons in premature infants. There is a need of further studies to understand the genetic background of BPD specific to different populations, to identify polymorphisms related with the disease and for developing genetic methods for early the diagnose of the disease.

With this purpose, first of all polymorphisms related with BPD and those which are related with similar other lung diseases will be investigated. DNA samples derived from blood samples of 200 patients (100 BPD infant and 100 control) will be examined for polymorphisms in specific genes that are chosen in the light of the prior literature scanning. To the investigators' knowledge, this will be the first study of a broad scanning of polymorphisms related with BPD in Turkish population.

ELIGIBILITY:
Inclusion Criteria:

* infants born under 30 gestational week
* infants with bronchopulmonary displasia

Exclusion Criteria:

* major congenital abnormalities
* lack of data
* parents don't agree with informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
DNA | 6 months
  Single nucleotide gene polymorphisms

CONTACTS AND LOCATIONS:
Overall Officials: Seda Yilmaz Semerci, Study Chair — Kanuni Sultan Suleyman Training and Research Hospital; Ayberk Akat, Principal Investigator — Istanbul Demiroglu Bilim University; Osman Mutluhan Ugurel, Study Chair — Yildiz Technical University; Merih Cetinkaya, Study Director — Kanuni Sultan Suleyman Training and Research Hospital; Dilek Turgut Balık, Study Director — Yildiz Technical University
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)

REFERENCES:
- [Derived] Akat A, Yilmaz Semerci S, Ugurel OM, Erdemir A, Danhaive O, Cetinkaya M, Turgut-Balik D. Bronchopulmonary dysplasia and wnt pathway-associated single nucleotide polymorphisms. Pediatr Res. 2022 Sep;92(3):888-898. doi: 10.1038/s41390-021-01851-6. Epub 2021 Dec 1. PMID 34853430